CLINICAL TRIAL: NCT00665860
Title: Safety, Efficacy, and Optimal Dosage of Soy Isoflavones to Prevent Osteoporosis
Brief Title: Safety and Effectiveness of Soy Phytoestrogens to Prevent Bone Loss
Acronym: OPUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: University of California (Other); Kaiser Foundation Research Institute (Other); University of Georgia (Other); University of Alabama at Birmingham (Other); Texas A&M University (Other)
Responsible Party: Principal Investigator, William Wong, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: TEXW-2001-04550; 2001-52102-11255
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Soy isoflavones; Postmenopausal women; Safety; Efficacy; Effective dosage
MeSH Terms: conditions — Osteoporosis | interventions — Soybean Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo
- 2 (Active Comparator)
  Interventions: Dietary Supplement: Soy isoflavones
- 3 (Active Comparator)
  Interventions: Dietary Supplement: Soy isoflavones

INTERVENTIONS:
Dietary Supplement: Placebo — Three pills per day for two years
  Arms: 1
Dietary Supplement: Soy isoflavones — Three pills that delivered 80 mg of aglycone isoflavones per day for two years
  Other Names: Soy germ isoflavones
  Arms: 2
Dietary Supplement: Soy isoflavones — Three pills that delivered 120 mg aglycone isoflavones per day for two years
  Other Names: Soy germ isoflavones
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether soy isoflavone supplementation is safe and effective to prevent bone loss in postmenopausal women.

DETAILED DESCRIPTION:
Over-the-counter soy isoflavone supplement usage is becoming common among postmenopausal women. However, there is no documented scientific evidence of its long-term safety and efficacy in preventing osteoporosis. Our primary goal is to determine the safety, efficacy, and optimal dosage of isoflavone supplementation to reduce bone loss in postmenopausal women. The multi-state, multi-institutional design ensures that the study results are representative of postmenopausal women in the U.S. population. Confirming the skeletal benefits of soy isoflavones could translate into reduced healthcare costs related to osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to swallow the pills
* No menses for 12 months
* Blood follicle stimulating hormone great than 30 IU/mL
* Lumbar spine bone mineral density t-score equal to or greater than -1.5

Exclusion Criteria:

* Strict vegetarians
* Current or recent smokers (within last five years)
* Abnormal screening mammogram, Pap smear and blood chemistries
* Clinical diagnosis of osteoporosis, spine and/or hip fracture, cancer, liver, kidney, gallbladder and heart disease
* Clinical diagnosis of psychiatric disorder
* Any allergic reactions to soy products
* Current treatment with bisphosphonates, calcitonin, fluoride, corticosteroids, tamoxifen, raloxifene, HRT, premarin, farestron and letrozole
* Current usage of black cohosh, blue cohosh, dong quai, Caltrate 600+Soy, Estroven, ginseng, Healthy Women, Natural Estrogen, Opti-Soy, PhytoFem, Probalance, Promensil, Remifemin, Rimostil and Trinovin

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 403 (Actual)
Dates: Start 2001-04; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | One year and two years

SECONDARY OUTCOMES:
Blood biochemical bone markers (osteocalcin, bone-specific alkaline phosphatase, cross-linked N-telopeptides of type 1 collagen) | One year and two years

CONTACTS AND LOCATIONS:
Overall Officials: William W. Wong, Ph.D., Study Director — Baylor College of Medicine
Locations (3):
- United States (3):
  - University of California, Davis, California
  - University of Georgia, Athens, Georgia
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Result] Ellis KJ, Shypailo RS, Steinberg FM, Lewis RD, Young RL, Wong WW. Reproducibility of fan-beam DXA measurements in adults and phantoms. J Clin Densitom. 2004 Winter;7(4):413-8. doi: 10.1385/jcd:7:4:413. PMID 15618602
- [Derived] Steinberg FM, Murray MJ, Lewis RD, Cramer MA, Amato P, Young RL, Barnes S, Konzelmann KL, Fischer JG, Ellis KJ, Shypailo RJ, Fraley JK, Smith EO, Wong WW. Clinical outcomes of a 2-y soy isoflavone supplementation in menopausal women. Am J Clin Nutr. 2011 Feb;93(2):356-67. doi: 10.3945/ajcn.110.008359. Epub 2010 Dec 22. PMID 21177797
- [Derived] Wong WW, Lewis RD, Steinberg FM, Murray MJ, Cramer MA, Amato P, Young RL, Barnes S, Ellis KJ, Shypailo RJ, Fraley JK, Konzelmann KL, Fischer JG, Smith EO. Soy isoflavone supplementation and bone mineral density in menopausal women: a 2-y multicenter clinical trial. Am J Clin Nutr. 2009 Nov;90(5):1433-9. doi: 10.3945/ajcn.2009.28001. Epub 2009 Sep 16. PMID 19759166